CLINICAL TRIAL: NCT04179825
Title: Integration of the Quick Parenting Assessment (QPA) Into Pediatrics: Parents and Clinicians' Perspectives
Brief Title: Parents' and Clinicians' Perspectives of the Quick Parenting Assessment (QPA)
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Seth Scholer, Professor, Vanderbilt University Medical Center
Other Study IDs: 180956
Record Dates: First submitted 2019-11-07; First posted 2019-11-27 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Social Stress; Parenting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A quality improvement (QI) study that integrates an adverse childhood experiences (ACEs) instrument, including the Quick Parenting Assessment (QPA), into pediatric primary care visit.

DETAILED DESCRIPTION:
Adverse childhood experiences (ACEs) are social determinants of health. ACEs include exposure to unhealthy parenting and family dysfunction. It is known that people who are exposed to adverse childhood experiences (ACEs) are at increased risk of over 40 health problems; some of these include heart disease, lung disease, obesity, smoking, alcoholism, illicit drug use, depression, suicide, and violence. The American Academy of Pediatrics recommends that primary care providers screen for and address ACEs/social determinants of health as part of the routine primary care visit.

Efforts are needed to develop and test algorithms that assess for ACEs in pediatric primary care and intervene as indicated.

The investigators have tested an ACEs screening instrument that includes the Quick Parenting Assessment with hundreds of parents of 2-10 year old children in the pediatric primary care clinic at Vanderbilt without incident (please see IRB# 161987).

The next step is a quality improvement (QI) study that integrates an ACEs screening algorithm into pediatric primary care visit.

In this study, the investigators integrate the Quick Parenting Assessment into the pediatric primary care visit at the 15 month, 30 month, 5 year, and 8 year visit. Key measures include parents' and health care providers' perspectives on the new service.

ELIGIBILITY:
Inclusion Criteria:

* Parents of 1-10 year old children presenting to a pediatric clinic for a well child visit.

Exclusion Criteria: Parents who do not speak English, Spanish, or Arabic.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents of young children presenting with their child for a well visit.
Sampling Method: Non-Probability Sample
Enrollment: 582 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Parent feedback | One day. The outcome will be assessed on same day as enrollment.
  Parents provide feedback regarding whether the new ACEs screening tool works for them using a questionnaire. The questionnaire included questions about whether the ACEs assessment worked for the parent and whether it was culturally sensitive.
Health care provider feedback. | One day. This outcome will be assessed on same day as the parent's enrollment.
  Health care providers provide feedback regarding whether the new ACEs screening tool works for them using a questionnaire. The questionnaire will include questions such as time spent reviewing the screening tool and whether the screening tool resulted in recommendations that would have otherwise not been made.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided